CLINICAL TRIAL: NCT02444663
Title: Validation of a Device for Performing Valgus and Varus Stress X-rays of the Knee
Brief Title: Validation of a Stress Device for the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Thomas Hamilton, Clinical Research Fellow, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 109367
Record Dates: First submitted 2015-04-27; First posted 2015-05-14 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will have the interventions in each of the ten arms of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Clinician Valgus (Active Comparator): Clinician performed fluoroscopic valgus and varus stress X-rays
  Interventions: Radiation: Clinician Valgus
- Clinician Varus (Active Comparator): Clinician performed fluoroscopic varus stress X-rays
  Interventions: Radiation: Clinician Varus
- Device Valgus - 0 Newton force (Experimental): Device performed fluoroscopic valgus stress X-rays - 0 Newton force
  Interventions: Radiation: Device Valgus - 0 Newton
- Device Valgus - 10 Newton force (Experimental): Device performed fluoroscopic valgus stress X-rays - 10 Newton force
  Interventions: Radiation: Device Valgus - 10 Newton
- Device Valgus - 20 Newton force (Experimental): Device performed fluoroscopic valgus stress X-rays - 20 Newton force
  Interventions: Radiation: Device Valgus - 20 Newton
- Device Valgus - 30 Newton force (Experimental): Device performed fluoroscopic valgus stress X-rays - 30 Newton force
  Interventions: Radiation: Device Valgus - 30 Newton
- Device Varus - 0 Newton force (Experimental): Device performed fluoroscopic varus stress X-rays - 0 Newton force
  Interventions: Radiation: Device Varus - 0 Newton
- Device Varus - 10 Newton force (Experimental): Device performed fluoroscopic varus stress X-rays - 10 Newton force
  Interventions: Radiation: Device Varus - 10 Newton
- Device Varus - 20 Newton force (Experimental): Device performed fluoroscopic varus stress X-rays - 20 Newton force
  Interventions: Radiation: Device Varus - 20 Newton
- Device Varus - 30 Newton force (Experimental): Device performed fluoroscopic varus stress X-rays - 30 Newton force
  Interventions: Radiation: Device Varus - 30 Newton

INTERVENTIONS:
Radiation: Clinician Valgus — Clinician performed valgus stress X-ray under fluoroscopy
  Arms: Clinician Valgus
Radiation: Clinician Varus — Clinician performed varus stress X-ray under fluoroscopy
  Arms: Clinician Varus
Radiation: Device Valgus - 0 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed valgus stress X-ray under fluoroscopy.
  Arms: Device Valgus - 0 Newton force
Radiation: Device Valgus - 10 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed varus stress X-ray under fluoroscopy.
  Arms: Device Valgus - 10 Newton force
Radiation: Device Valgus - 20 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed valgus stress X-ray under fluoroscopy.
  Arms: Device Valgus - 20 Newton force
Radiation: Device Valgus - 30 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed valgus stress X-ray under fluoroscopy.
  Arms: Device Valgus - 30 Newton force
Radiation: Device Varus - 0 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed valgus stress X-ray under fluoroscopy.
  Arms: Device Varus - 0 Newton force
Radiation: Device Varus - 10 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed valgus stress X-ray under fluoroscopy.
  Arms: Device Varus - 10 Newton force
Radiation: Device Varus - 20 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed valgus stress X-ray under fluoroscopy.
  Arms: Device Varus - 20 Newton force
Radiation: Device Varus - 30 Newton — Device (Oxford Stress System for Knee Arthroplasty Radiographs (OSSKAR)) performed valgus stress X-ray under fluoroscopy.
  Arms: Device Varus - 30 Newton force

SUMMARY:
X-rays are the most frequently used imaging test when evaluating the knee for joint replacement. They are non-invasive, safe and cost effective. They allow assessment of: progression of disease, appropriateness for joint replacement (in particular unicompartmental knee replacement (UKR)) as well as likely prognosis following replacement.

Currently standard assessment involves: standing anteroposterior, lateral and skyline X-ray views. In addition in patients being considered for joint replacement valgus/varus stress X-rays are used to evaluate the lateral compartment (as well as medial collateral ligament) and medial compartment respectively to assess the status of the cartilage. Stress X-rays require the clinician to attend X-ray, often during busy clinics, exposing them to additional radiation, and as such they are seldom performed.

A patient and user friendly device for performing valgus and varus stress X-rays of the knee for diagnostic and pre-operative planning purposes in the setting of knee replacement surgery has been developed. This device has the potential to benefit patients as it will allow an accurate assessment of the pattern and severity of arthritis affecting their knee without the need for additional diagnostics such as MRI or arthroscopy. Furthermore for healthcare practitioners and providers this device will facilitate the smooth running of clinics and reduce the additional clinic appointments required to review MRI results. Ultimately this device will allow an informed discussion about treatment options, reduce the pre-operative uncertainty about suitability for UKR in those undergoing surgery and ensure that those patients who are suitable for UKR benefit from this procedure. This device will help ensure that patients receive the optimum treatment in a clinically and cost efficient manner.

This study will validate valgus and varus stress X-rays performed using the investigators' device against the gold standard of clinician performed manual stress.

DETAILED DESCRIPTION:
X-rays are the most frequently used imaging test when evaluating the knee for joint replacement. They are non-invasive, safe and cost effective. They allow assessment of: progression of disease, appropriateness for joint replacement (in particular unicompartmental knee replacement (UKR)) as well as likely prognosis following replacement.

Currently standard assessment involves: standing anteroposterior, lateral and skyline X-ray views. In addition in patients being considered for joint replacement valgus/varus stress X-rays are used to evaluate the lateral compartment (as well as medial collateral ligament) and medial compartment respectively to assess the status of the cartilage.

The assessment of pattern and severity of disease is critical when evaluating suitability for joint replacement and well as when deciding between total knee replacement (TKR), where all articulating surface are replaced, or UKR, where only the diseased portion of the joint is replaced. Understanding the pattern of disease is essential to ensure appropriate patient selection for UKR, which is appropriate in up to half of patients undergoing knee replacement, and has significant benefits over TKR including: half the risk of venous thromboembolism, myocardial infarction or deep infection, two thirds the risk of stroke, one quarter the risk of blood transfusion and significantly lower mortality up to eight years following their operation.

Stress X-rays are currently performed by the clinician, requiring them to attend radiology, often during clinic. To perform the stress views the clinician fixes the knee and moves the tibia away from the midline, valgus stress, where an X-ray is taken. The alignment of this view is confirmed before the tibia is moved towards the midline, varus stress, where another X-ray is taken. Stress X-rays are resource dependent and can be time consuming. In addition, the technique can be uncomfortable for patients as well as resulting in additional radiation exposure to the clinical practitioner. On an average, a knee surgeon may be exposing themselves to excess of 300 exposures every year with the cumulative effect of radiation exposure being significant. As such in many centers stress views are often not performed, and as standing antero-posterior X-ray views are inadequate to assess disease severity and pattern many clinicians have adopted additional imaging modalities such as MRI or direct observation via arthroscopy to evaluate the status of the cartilage in each compartment. The use of these additional imaging techniques introduces significant additional costs as well as delays to treatment. Furthermore the long term outcomes of UKR have been established using stress views, and as a consequence outcomes based on MRI or arthroscopic findings have not been fully established.

A patient and user friendly device for performing valgus and varus stress X-rays of the knee for diagnostic and pre-operative planning purposes in the setting of knee replacement surgery has been developed. This device has the potential to benefit patients as it will allow an accurate assessment of the pattern and severity of arthritis affecting their knee without the need for additional diagnostics such as MRI or arthroscopy. Furthermore for healthcare practitioners and providers this device will facilitate the smooth running of clinics and reduce the additional clinic appointments required to review MRI results. Ultimately this device will allow an informed discussion about treatment options, reduce the pre-operative uncertainty about suitability for UKR in those undergoing surgery and ensure that those patients who are suitable for UKR benefit from this procedure. This device will help ensure that patients receive the optimum treatment in a clinically and cost efficient manner.

This study will validate valgus and varus stress X-rays performed using the investigators' device against the gold standard of clinician performed manual stress.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 50 years or above.
* Knee osteoarthritis any grade, affecting the tibio-femoral joint
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Previous joint replacement on ipsilateral knee
* Previous anterior cruciate ligament reconstruction or injury
* Previous high tibial osteotomy
* Previous intra-articular fracture
* History of Inflammatory arthritis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

REFERENCES:
- See also: Oxford Orthopaedic Engineering Centre, Nuffield Department of Orthopaedics, Rheumatology and Musculoskeletal Sciences (NDORMS), University of Oxford — https://www.ndorms.ox.ac.uk/research-groups/oxford-orthopaedic-engineering-centre

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 9 participants recruited with the interventions in each arm applied to all participants
Groups:
- All Study Participants: All study participants Clinician Valgus Clinician Varus Device Valgus 0N Device Valgus 10N Device Valgus 20N Device Valgus 30N Device Varus 0N Device Varus 10N Device Varus 20N Device Varus 30N
Period: Clinician Valgus
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Clinician Varus
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Valgus 0N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Valgus 10N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Valgus 20N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Valgus 30N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Varus 0N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Varus 10N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Varus 20N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Device Varus 30N
Arm/Group | All Study Participants
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 70 [63 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9

OUTCOME MEASURES:

1. Primary Outcome: Compartment Specific Knee Minimum Joint Space Width (Varus - Medial Compartment, Valgus - Lateral Compartment)
Description: Knee minimum joint space width measured on anteroposterior fluoroscopic images using custom, validated, in house software (KneeMorph, MATLAB, MathWorks, Massachusetts).
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Clinician Valgus | Clinician Varus | Device Valgus - 0 Newton Force | Device Valgus - 10 Newton Force | Device Valgus - 20 Newton Force | Device Valgus - 30 Newton Force | Device Varus - 0 Newton Force | Device Varus - 10 Newton Force | Device Varus - 20 Newton Force | Device Varus - 30 Newton Force
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
mm | 7.42 (1.38) | 3.92 (2.12) | 8.22 (1.3) | 7.47 (1.54) | 7.31 (1.71) | 7.33 (1.62) | 8.56 (1.44) | 4.41 (1.83) | 3.7 (2.08) | 3.84 (2.28)

2. Secondary Outcome: Pain (VAS 0 - 10)
Description: Pain Score during stress radiographs (VAS 0 - 10) where a higher score represents more pain (10 = worst pain).
Time Frame: At time of procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinician Valgus | Clinician Varus | Device Valgus - 0 Newton Force | Device Valgus - 10 Newton Force | Device Valgus - 20 Newton Force | Device Valgus - 30 Newton Force | Device Varus - 0 Newton Force | Device Varus - 10 Newton Force | Device Varus - 20 Newton Force | Device Varus - 30 Newton Force
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale | 3.67 (2.08) | 4.00 (2.00) | 0 (0) | 0.78 (0.74) | 1.56 (2.35) | 5.44 (2.01) | 0 (0) | 0.88 (1.64) | 1.25 (2.31) | 4.88 (1.36)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Clinician Valgus | Clinician Varus | Device Valgus - 0 Newton Force | Device Valgus - 10 Newton Force | Device Valgus - 20 Newton Force | Device Valgus - 30 Newton Force | Device Varus - 0 Newton Force | Device Varus - 10 Newton Force | Device Varus - 20 Newton Force | Device Varus - 30 Newton Force
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes